CLINICAL TRIAL: NCT00302094
Title: Image Fusion PET, CT and 3D-ultrasound Examinations in Treatment of Anal Cancer
Brief Title: Image Fusion PET, CT and 3D-ultrasound Examinations
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Caroline Ewertsen, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: (KF) 11-107/03
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
CT-examinations are used in computer programs which are used in the planning of external radiation of cancers in the anal canal. In CT the structures of the anal canal are hardly visible. 3D-ultrasound examinations offer a better visualisation of normal and pathological structures of the anal canal. The description of the tumour made from the 3D-ultrasound examination is used in the planning of the external radiation.

PET-CT is used to visualise tumour activity also in lymp nodes. The hypothesis of the study is that image fusion of PET, CT and 3D-ultrasound will offer better visualisation of tumour and hereby more accurate diagnostics and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified cancer of the anal canal

Exclusion Criteria:

* Pregnancy
* Unability to cooperate to radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anal cancer
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Program to fuse 3D ultrasound and PET/CT data | april 2009

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Nielsen, Dmsci, phd., Study Director — Rigshospitalet, Denmark; Caroline Ewertsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Clinic of Radiology, Section of Ultrasound, Rigshospitalet, Copenhagen, Denmark